CLINICAL TRIAL: NCT02359201
Title: Double-blind, Randomized, Placebo-controlled, Cross-over Study of the Effect of a 1.5 mg Nicotine Lozenge on Smoking Craving
Brief Title: Assessment of V0018 1.5 mg Effect on Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V00018 PC 2 07; 2014-004424-21 (EudraCT Number)
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Smoking
Keywords: Nicotine replacement therapy; craving; Healthy moderately dependant smokers
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sequence 1 (Experimental): Treatment group sequence: Test Product (V0018) on Day 1 and Placebo on Day 2
  Interventions: Drug: V0018; Drug: Placebo
- Sequence 2 (Experimental): Treatment group sequence: Placebo on Day 1 and Test Product (V0018) on Day 2
  Interventions: Drug: V0018; Drug: Placebo

INTERVENTIONS:
Drug: V0018 — Oromucosal - Single dose
Drug: Placebo — Oromucosal - Single dose

SUMMARY:
The purpose of this study is to evaluate the reduction of craving after administration of V0018 1.5 mg compared to placebo in healthy moderately dependent smokers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 to 64 years
* Smoking ≥ 10 cigarettes/day and < 20 cigarettes/day continuously for the last two years
* With a first cigarette smoked within 30 min after waking
* Not currently in the process of quitting smoking

Exclusion Criteria:

Related to pathologies

* Current or recurrent buccal lesions which, in the opinion of the investigator, would interfere with the assessment of the different parameters
* Hyposalivation or asialia
* Intolerance to lactose, or any pathology that could cause endogenous production of Carbon Monoxide (CO)

Related to treatments

* Use of antidepressants within the last three months
* Use of sedatives, hypnotics, tranquilizers or any other addictive agents within the last 3 months
* Routine use of tobacco other than cigarettes
* Regular use for more than one week of any treatment for smoking cessation (gum, patch, inhaler, lozenge, tablet, bupropion, varenicline) and other smokeless tobacco products (including e-cigarettes) within three months
* History of hypersensitivity to nicotine, peanut, soya or to any of the excipients of study treatment
* Intolerance to fructose
* History of phenylketonuria (aspartame)

For women of childbearing potential:

* Is pregnant or in post-partum period or a nursing mother

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Questionnaire for Smoking Urges Brief (QSU-Brief) (10 items) | 15 minutes
  Change from study baseline to 15 minutes after treatment intake for the QSU-brief total score and demonstrate any earlier effect.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise MD TONNER, Study Director — Pierre Fabre Medicament
Locations (1):
- Gières, France